CLINICAL TRIAL: NCT05437081
Title: A Family-Based Alcohol Preventive Intervention for Latino Emerging Adults
Acronym: LEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06162016.026
Record Dates: First submitted 2021-11-30; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Binge Alcohol Consumption; Risk Behavior, Health; Driving Under the Influence; High-Risk Sex; Identity, Social; Parenting
MeSH Terms: conditions — Binge Drinking; Health Risk Behaviors; Driving Under the Influence; Unsafe Sex; Social Identification

STUDY DESIGN:
Intervention Model Description: Latino emerging adults (EAs)and Latino parents of EAs were recruited in Oregon and Florida. Participants were then randomly selected into either the intervention or the control condition. Participants randomized to the control condition received referrals to community agencies for mental health, substance abuse, and health issues commonly experienced by EAs. Participants randomized to the intervention condition were invited to attend four family-focused sessions (for parents) or four identity development-focused sessions (for EAs).
Who Masked: Outcomes Assessor
Masking Description: Though most assessments were conducted by participants themselves online, in a few cases, study assessors conducted telephone interviews with parent participants. In these cases, the assessor was kept blind to the participant's study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMERGE program (Experimental): Participants were randomly assigned to one of two conditions: intervention or control. Intervention participants engaged in a 4 session program named the EMERGE program focused on identity development (emerging adults) or support for emerging adults (parents). Control participants received referrals to community agencies for behavioral and mental health support as needed.
  Interventions: Behavioral: Latino Emerging Adults (LEA)
- Referral services as needed (No Intervention): Participants were randomly assigned to one of two conditions: intervention or control. Control participants received services as usual.

INTERVENTIONS:
Behavioral: Latino Emerging Adults (LEA) — The LEA program involves two components, one for emerging adults (aged 18-23 years old) focused on identity development linked to cultural and familial strengths, and a parent component focused on support for emerging adult children. Each session is 4 sessions.
  Arms: EMERGE program

SUMMARY:
The purpose of the proposed study was to develop a family-based drinking prevention intervention for Latino emerging adults (EAs) and Latino parents of EAs. Although drinking rates for Latinos are lower than those for Whites in terms of the prevalence of alcohol use, the consequences of alcohol use (e.g., drunk driving, unplanned/unprotected sex, alcohol-related injuries) appear to be more severe for Latinos, especially those 18-23 years old. The investigators developed a brief (4 session) intervention for each of EAs and parents focused on identity development and parent support for EAs, respectively.

DETAILED DESCRIPTION:
The purpose of the proposed study was to develop a family-based drinking prevention intervention for Latino emerging adults (EAs) and Latino parents of EAs. The investigators specifically targeted EAs aged 18-23. Although drinking rates for Latinos are lower than those for Whites in terms of the prevalence of alcohol use, the consequences of alcohol use (e.g., drunk driving, unplanned/unprotected sex, alcohol-related injuries) appear to be more severe for Latinos, especially those 18-23 years old.

The intervention program included four sessions with emerging adults (EA) in a group setting, and four sessions with groups of parents of EAs. This dual-site project was developed in Oregon and Florida in three phases: (1) development of the intervention components; (2) initial pilot testing and focus group feedback (including modifying the intervention and revising the manuals); and (3) a randomized pilot study. The EA component was developed by integrating identity-based intervention strategies that have been used successfully with adolescents and EAs, ensuring that they are developmentally and culturally appropriate. The parenting component was developed by adapting efficacious parenting strategies used with adolescents so that the activities were developmentally and culturally appropriate for parents of EAs. As the pilot study launch coincided with the start of the COVID-19 pandemic, the investigators adapted the original in-person approaches for online delivery.

ELIGIBILITY:
Inclusion criteria:

Emerging adult criteria:

* Between the ages of 18 and 23 years old upon recruitment
* Identify as Latina/o, Hispanic, Chicana/o, or have been born or descended from a parent or grandparent from Mexico or another nation in Central or South America or the Spanish-speaking Caribbean
* Intend to remain in the area for the four months following their recruitment into the study in order to participate in the intervention, if selected

Parent criteria:

* Have a child between the ages of 18 and 23 years old
* Identify as Latina/o, Hispanic, Chicana/o, or have been born or descended from a parent from Mexico, or a nation in Central or South America or the Spanish-speaking Caribbean
* Speak and understand Spanish

Exclusion Criteria:

Emerging adult criteria:

• EAs are not themselves a parent or stepparent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Emerging Adult Self-Efficacy | 3-4 months
  The Latino Emerging Adult (LEA) Self-Efficacy scale was designed to appraise Latino emerging adults' healthy identity formation and healthy behaviors. Participating emerging adults self-administered this online assessment twice during the study--at baseline, pre-intervention, and 3-4 months post-intervention. The scale includes 14 items (e.g., I feel confident that I can successfully tackle the challenges of becoming an adult; I draw on strengths from my family's cultural background to help me deal with the stress of becoming an adult; I use healthy activities to deal with stress; Mentors [parents or other trusted adults] are important in the life success of emerging adults). Answer choices include: 1-Strongly disagree; 2-Disagree; 3-Agree; 4-Strongly Agree. Higher scores indicate higher emerging adult self-efficacy. The Cronbach's alpha was .78. (Citation: Center for Equity Promotion. [2019]. Latino Emerging Adult Self-Efficacy scale. University of Oregon.)
Parent-Emerging Adult Relationship Quality | 3-4 months
  The Latino Emerging Adult (LEA) Parent-Emerging Adult Relationship Quality scale was designed by the research team. Participating emerging adults self-administered this online computer-based survey twice during the study--at baseline and approximately 3-4 months later, after the completion of the intervention program. The scale includes 6 items (e.g., Even though my parent can be annoying, I know that she/he is my best supporter; Even when I think that my parent is wrong, I understand where she/he is coming from). Answer choices include: 0-Not at all true; 1-Not really true; 2-Somewhat true; 3-Very true. Higher scores equal higher quality relationships as reported by emerging adults. The Cronbach's alpha was .82. (Citation: Center for Equity Promotion. [2019]. Latino Emerging Adult Parent-Emerging Adult Relationship Quality scale. University of Oregon.)
Parent Trust in Emerging Adult Decision-Making | 3-4 months
  The Latino Emerging Adult (LEA) Parent Trust in Emerging Adult Decision-Making scale was designed by the research team. Participating parents self-administered this online computer-based survey twice during the study--at baseline and approximately 3-4 months later, after the completion of the intervention program. The scale includes 6 items (e.g., I am confident that my emerging adult child will make the right choices in life; I'm afraid that my emerging adult child will not be able to figure out what to do in life; My emerging adult child knows what to do when s/he needs to make an important life decision). Answer choices include: 0-Not at all true; 1-Not really true; 2-Somewhat true; 3-Very true. Higher scores indicate higher parent-reported trust in emerging adult children's decision-making. The Cronbach's alpha was .77. (Citation: Center for Equity Promotion. [2019]. Latino Emerging Adult (LEA) Parent Trust in Emerging Adult Decision-Making scale. University of Oregon.)
Parent support | 3-4 months
  The Latino Emerging Adult (LEA) Parent Support scale was designed by the research team. Participating parents self-administered this online computer-based survey twice during the study--at baseline and approximately 3-4 months later, after the completion of the intervention program. The scale includes 8 items (e.g., Even if [child's name] doesn't listen to me one time, I still know that I can get through to him/her the next time; [child's name] comes to me and talks to me about important issues in his/her life; I generally know how to connect with or reach out to [child's name] when they need my support). Answer choices include: 1-Strongly disagree; 2-Disagree; 3-Agree; 4-Strongly Agree. Higher scores indicate higher parent support. The Cronbach's alpha was .82. (Citation: Center for Equity Promotion. [2019]. Latino Emerging Adult (LEA) Parent Support scale. University of Oregon.)
Emerging adult alcohol consumption | 3-4 months
  Three items from the University of Michigan's Monitoring the Future survey were used to appraise alcohol use (Johnston, L. D., O'Malley, P. M., Bachman, J. G., Schulenberg, J. E., & Miech, R. A. (2015). Monitoring the Future national survey results on drug use, 1975-2014: Volume II, college students and adults ages 19-55.). Items include:
  1. Have ever tried even a few sips of alcohol? Yes No (if no, skip to #3)
  2. If YES: How old were you when you first tried at least a few sips of alcohol? _____ years old
  3. During the last 3 months, what was the HIGHEST number of drinks that you drank in a single day?
Drinking-related risk behaviors | 3-4 months
  Twelve items from the Monitoring the Future survey were used (Johnston, L. D., O'Malley, P. M., Bachman, J. G., Schulenberg, J. E., & Miech, R. A. (2015). Monitoring the Future national survey results on drug use, 1975-2014: Volume II, college students and adults ages 19-55). Exemplar items include: During the last 3 months, about how many days did you drink until it affected your ability to make decisions?; How many times in the last 3 months did you use other drugs after you had been drinking?; and, In the past 3 months, how many times did you ride in a car when you knew the driver was drunk or high?
Drinking-related harm reduction behaviors | 3-4 months
  The Latino Emerging Adult (LEA) Drinking-related Harm Reduction Behaviors scale was designed by the research team. Participating emerging adults self-administered this online survey twice during the study--at baseline and approximately 3-4 months later, after the completion of the intervention program. The scale includes 13 items (e.g., If one of my friends is really drunk, I make sure that person is safe; If I have been drinking too much I feel comfortable finding a ride home with a sober driver or finding a place to sleep; In my group of friends, if someone has been drinking too much we make sure that he/she doesn't drive). Answer choices include: 1-Strongly disagree; 2-Disagree; 3-Agree; 4-Strongly Agree. Higher scores indicate EAs practice more alcohol-related harm-reducing behaviors. The Cronbach's alpha was .93. (Citation: Center for Equity Promotion. [2019]. Latino Emerging Adult (LEA) Drinking-related Harm Reduction Behaviors scale. University of Oregon.)
Emerging adult perceived stress | 3-4 months
  Emerging adult participants respond in an online survey to the 10-item Perceived Stress Scale (PSS-10; Cohen, S. and Williamson, G. [1988]. Perceived stress in a probability sample of the United States. In S. Spacapan & S. Oskamp [Eds.] The social psychology of health [pp. 31-67]. Sage Publications, Inc.). Answer choices range from Never = 0 to Very often = 4. Responses are summed with higher sum scores reflecting higher perceived stress. The Cronbach's alpha for emerging adults in this study was .82.
Parent perceived stress | 3-4 months
  Parent participants respond in an online survey to the 10-item Perceived Stress Scale (PSS-10; Cohen, S. and Williamson, G. [1988]. Perceived stress in a probability sample of the United States. In S. Spacapan & S. Oskamp [Eds.] The social psychology of health [pp. 31-67]. Sage Publications, Inc.). Answer choices range from Never = 0 to Very often = 4. Responses are summed with higher sum scores reflecting higher perceived stress.
Bicultural identity integration | 3-4 months
  Sixteen items from the Bicultural Identity Integration Scale (BIIS-2) were used to capture variation in emerging adults' experiences of acculturation. (Huynh, Q. L., Benet-Martínez, V., & Nguyen, A. M. D. [2018]. Measuring variations in bicultural identity across US ethnic and generational groups: Development and validation of the Bicultural Identity Integration Scale-Version 2 [BIIS-2]. Psychological Assessment, 30[12], 1581.). Exemplar items include: I feel part of a combined culture that is a mixture of Hispanic/Latino and American; I find it difficult to combine Hispanic/Latino and American cultures; I do not blend my Hispanic/Latino and American cultures. Answer choices range from 1 (strongly disagree) to 5 (Strongly agree). The scale taps cultural blendedness versus compartmentalization and cultural harmony versus conflict, and final scores are averages.
Emerging adult future orientation | 3-4 months
  Ten items from the Steinberg et al. Future Orientation Scale were used (Steinberg L, Graham S, O'Brien L, Woolard J, Cauffman E, Banich M. [2009]. Age differences in future orientation and delay discounting. Child Development. Jan-Feb;80[1]:28-44.) The 10 items include question numbers 2, 3, 4, 5, 7, 9, 10, 12, 13, 15 across 4 sub-scales including Planning Ahead, Time Perspective, Anticipation of Future Consequences, and Anticipation of Future Consequences. All items are scored left to right on a scale of 1-4. Reverse score items 1, 3, 4, 6, 8, 11, and 14, so that higher scores indicate a stronger future orientation.
Parent hope for emerging adult child's future | 3-4 months
  This 12 item scale appraises parents' hopes for their emerging adult children's future. Answer options range from 0-Not at all true to 3-Very true. Exemplar items include: It's important to me that (my child) continues her/his education after high school; It's important to me that (my child) graduates from college; I know what (my child's) goals are for her/his future; and I help (my child) make plans and take steps towards her/his goals for the future. Citation: Center for Equity Promotion. [2019]. Latino Emerging Adult (LEA) Parent Hope for Emerging Adult Future scale. University of Oregon.)
American identity integration | 3-4 months
  Seven items were used from the American Identity Measure (Schwartz et al [2012]. The American Identity Measure: Development and validation across ethnic subgroup and immigrant generation. Identity: An International Journal of Theory and Research, 12[2], 93-128.). Exemplar items include: I am happy that I am an American; I have a strong sense of belonging to the United States. Answer choices range from 1 (strongly disagree) to 5 (Strongly agree). Higher scores indicate higher American identity affirmation.

SECONDARY OUTCOMES:
Emerging adult acculturative stress | 3-4 months
  Items from the Multidimensional Acculturative Stress Inventory for Adults of Mexican Origin (MASI) were used (Rodriguez et al. [2002]. Development of the Multidimensional Acculturative Stress Inventory for Adults of Mexican Origin. Psychological Assessment, 14[4], 451-461.) The MASI is a 36-item stress measure that assesses acculturative stress among persons of Mexican origin living in the United States;10 items were selected that are part of factor 3: pressure to acculturate, and factor 4: pressure against acculturation. Response options begin with a stem: Has this occurred in the last 3 months? Yes or no. If yes, how worrying/stressful has this been? Follow-up response options range from 1-Not at all worrying/stressful to 5-Extremely worrying/stressful. Final scores reflect incidence of stress exposure (sum of "yes" stem responses) and stress responsiveness (average of follow-up stressfulness scores).
Parent acculturative stress | 3-4 months
  Items from the Multidimensional Acculturative Stress Inventory for Adults of Mexican Origin (MASI) were used (Rodriguez et al. [2002]. Development of the Multidimensional Acculturative Stress Inventory for Adults of Mexican Origin. Psychological Assessment, 14[4], 451-461.) The MASI is a 36-item stress measure that assesses acculturative stress among persons of Mexican origin living in the United States;10 items were selected that are part of factor 3: pressure to acculturate, and factor 4: pressure against acculturation. Response options begin with a stem: Has this occurred in the last 3 months? Yes or no. If yes, how worrying/stressful has this been? Follow-up response options range from 1-Not at all worrying/stressful to 5-Extremely worrying/stressful. Final scores reflect incidence of stress exposure (sum of "yes" stem responses) and stress responsiveness (average of follow-up stressfulness scores).

CONTACTS AND LOCATIONS:
Overall Officials: Heather H McClure, PhD, Principal Investigator — University of Oregon; Seth J Schwartz, PhD, Principal Investigator — University of Texas at Austin

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set is available to other researchers and can be accessed through contacting either study PI.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available by January 2022 and available indefinitely.
Access Criteria: Researchers interested in accessing the data must share their contact information with PIs.